CLINICAL TRIAL: NCT01262768
Title: Exploring the Accuracy and Acceptability of Portion Size Measurement Aids in Parents of Overweight Children
Brief Title: Efficacy of Portion Size Measurement Aids
Acronym: PSMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Geoff Ball, Associate Professor, Dept Pediatrics and Director, Pediatric Centre for Weight and Health, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00010835
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Nutrition Assessment; Obesity
Keywords: Nutrition; Obesity; Parent; Portion Size Estimation; Accuracy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2D Portion Size Measurment Aids (PSMAs) (Experimental): The 2D PSMAs are life-size photographs of the 3D PSMAs.
  Interventions: Behavioral: Portion Size Measurement Aids (PSMAs)
- 3D Portion Size Measurement Aids (PSMAs) (Experimental): The 3D PSMAs include foam rubber replicas of a golf ball, a hockey puck, a tennis ball and a baseball.
  Interventions: Behavioral: Portion Size Measurement Aids (PSMAs)

INTERVENTIONS:
Behavioral: Portion Size Measurement Aids (PSMAs) — Subjects are randomly assigned to receive either 2D or 3D PSMAs to examine accuracy, acceptability and usefulness of the models. Both groups receive brief instructions on the use of the respective PSMAs, complete an accuracy estimation task, and are given the 2D or 3D PSMAs to take home with them to use for 2-4 weeks, after which the researchers telephone parents to complete a brief satisfaction and usefulness survey.
  Other Names: 2D Portion Size Measurement Aids (PSMAs); 3D Portion Size Measurement Aids (PSMAs)

SUMMARY:
Portion size measurement aids (PSMAs) are tools that facilitate the estimation of food servings. The objectives of this study are to determine (a) if food portion size estimation accuracy differs when using a two dimensional (2D) PSMA (actual-size photos called Portion Size Cards) compared to a 3D PSMA (Portion Size Kit) and (b) whether differences exist in the short-term usefulness of and satisfaction with these PSMAs in a sample of parents of overweight children and youth. We hypothesize that the group that receives the 3D PSMAs will be more accurate in food portion size estimation and will be more satisfied with the tool compared to the group that receives the 2D PSMAs.

DETAILED DESCRIPTION:
Forty primary caregivers of overweight children and youth attending the Pediatric Centre for Weight and Health (Edmonton, AB) will be recruited. Participants will be randomly assigned to one of the two groups (2D PSMAs versus 3D PSMAs). After a brief explanation of the respective tool, participants will estimate the volumes of pre-measured rubber food portion models on a test plate. Participants will then be given the 2D or 3D PSMAs to take home with them to use in the real-world. After 2-4 weeks, participants will be telephoned by the research team to complete a brief survey to evaluate their usefulness of and satisfaction with the 2D or 3D PSMAs at home.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be primary caregivers of children or youth attending a clinical appointment for weight management (clients must have a BMI greater or equal to the 85th percentile at this clinic)
* Participants must be literate and fluent in English

Exclusion Criteria:

* Any participant who does not meet the above criteria
* Participants must not have had any previous education or resources on food portion sizes at this clinic

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-04; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of food portion size estimation | At the time of subject interview (single time point)
  During the initial interview, the subject receives a brief description of the task and is shown pre-estimated rubber food models. The subject then estimates the portion sizes (volumes) of the rubber food models using either 2D or 3D PSMAs.

SECONDARY OUTCOMES:
Acceptability (satisfaction and usefulness) of 2D and 3D PSMAs | 2-4 weeks following the accuracy assessment
  After the intial interview, subjects are given either 2D or 3D PSMAs to take home with them to use in a real-world setting. After 2-4 weeks, the researcher team contacts the subjects to complete a brief telephone interview to determine parental satisfaction and usefulness regarding the 2D or 3D PSMAs.

CONTACTS AND LOCATIONS:
Overall Officials: Geoff DC Ball, PhD, RD, Principal Investigator — Department of Pediatrics, University of Alberta; Director, Pediatric Centre for Weight and Health
Locations (1):
- Pediatric Centre for Weight and Health- Edmonton General Continuing Care Centre, Edmonton, Alberta, Canada